CLINICAL TRIAL: NCT06943105
Title: Effectiveness of Group-based Nonviolent Communication Interventions for Improving Mental Well-being in Parents: a Randomised Controlled Trial
Brief Title: Nonviolent Communication for Parents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Responsible Party: Principal Investigator, Dr Grace SUN Yuying, Assistant Professor, Hong Kong Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HE-RGC2024/NHS02
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Anxiety; Depression Symptom; Well-being
Keywords: Nonviolent Communication; parents; Depressive Symptoms; Anxiety
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Receiving NVC Interventions (Experimental): Participants in the intervention group will receive six weekly 1.5-hour face-to-face NVC training sessions delivered by trained social workers.
  Interventions: Behavioral: Nonviolent Communication Intervention
- Wailist Control Group (No Intervention): The waitlist control group will not receive any training before all the assessments have been done by both groups. The wailist control group will receive NVC training sessions after all assessments. During the whole study period, these participants can access usual medical services, whether related or unrelated to mental health needs.

INTERVENTIONS:
Behavioral: Nonviolent Communication Intervention — The intervention will be conducted by social workers who will be trained by professional NVC trainers through a train-the-trainer workshop, including six sessions. The interventions include an introduction to four fundamental principles of NVC, distinguishing observations from evaluations, identifying and expressing feelings, taking responsibility for feelings and needs, and using positive action language to make requests. Each session will feature a review of the previous session, a warm-up game and an exercise to consolidate the learning of the concepts. The intervention sessions will also include group discussions and debriefing sessions on parents' experiences of practising NVC.
  Arms: Receiving NVC Interventions

SUMMARY:
This randomised controlled trial (RCT) aims to evaluate the effectiveness of face-to-face Nonviolent Communication (NVC) intervention in improving parents' mental well-being and NVC skills, reducing parenting stress, depression and anxiety symptoms, and child emotional and behavioural problems.

A total of 172 parents with primary-school-age children will be recruited and randomly assigned to an intervention group or a waitlist control group. The intervention group will receive six weekly 1.5-hour face-to-face NVC training sessions delivered by trained social workers.

Five to ten social workers will be trained by professional NVC trainers through a train-the-trainer workshop, including three sessions. Each social worker will be assessed before (TTT1), after (TTT2) the workshops and 10 months (TTT3).

Assessments for participants will be conducted at baseline (T1), immediately post-intervention (T2), and at three-month follow-up (T3). After completing the assessments, the waitlist control group will receive the same sessions. Qualitative interviews will be conducted to explore participants' experiences and perceptions of NVC.

ELIGIBILITY:
Inclusion Criteria:

* 1) parents aged 24-59 years with children of primary school age;
* 2) with mild to severe depressive symptoms (score >5 on the Patient Health Questionnaire (PHQ)-9) (Kroenke et al., 2001) and/or mild to severe anxiety symptoms (score >5 on the General Anxiety Disorder (GAD)-7) (Spitzer et al., 2006); and
* 3) Hong Kong residents who can understand Cantonese.

Exclusion Criteria:

* 1) under psychiatric treatment, psychotherapy groups and are classified as unstable cases based on the judgment of the recruiting social workers;
* 2) participating in other related parenting programmes.

Ages: 24 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 172 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Well-being | T1: Baseline; T2: Immediate post-intervention; T3: 3 months post-T2
  The Short Warwick-Edinburgh Mental Well-being Scale (SWEMWS) is a 7-item scale for assessing mental health in non-clinical populations. Using a 5-point Likert scale (1 = none of the time, 5 = all the time), the total score is calculated by summing all seven items. The Chinese version showed good validity and reliability in the investigators' previous study. The congeneric reliability was 0.85 and the test-retest reliability was 0.70.
NVC skills | T1: Baseline; T2: Immediate post-intervention; T3: 3 months post-T2
  The measure of NVC skills was developed based on a 16-item scale that represents the four principles of NVC skills. Each item is rated on a 5-point scale ranging from 0 = never to 5 = always. The average score is calculated, with higher scores indicating better NVC skills. Cronbach's alpha was 0.82 in the investigators' pilot study.

SECONDARY OUTCOMES:
Parenting stress | T1: Baseline; T2: Immediate post-intervention; T3: 3 months post-T2
  The Parental Stress Scale (PSS) is an 18-item questionnaire that assesses feelings about parents' parenting role. A 16-item version of the PSS was developed by Leung et al. for Hong Kong parents. Responses are given on a 5-point scale. The Chinese version showed good internal consistency (Cronbach's alpha: 0.86).
Depressive symptoms | T1: Baseline; T2: Immediate post-intervention; T3: 3 months post-T2
  The Patient Health Questionnaire (PHQ)-9 is a 9-item instrument that is commonly used to measure depressive symptoms in the past two weeks. Each item is rated on a 4-point scale ranging from 0 = not at all to 3 = nearly every day. The Chinese version showed good validity and reliability (Cronbach's alphas: 0.82-0.92).
Anxiety | T1: Baseline; T2: Immediate post-intervention; T3: 3 months post-T2
  The Generalized Anxiety Disorder (GAD)-7 scale is a 7-item instrument to assess generalised anxiety disorder in the past two weeks. The response options for the seven symptoms are the same as PHQ-9. The Chinese version showed good validity and reliability (Cronbach's alphas: 0.89-0.95).
Child emotional and behavioural problems | T1: Baseline; T2: Immediate post-intervention; T3: 3 months post-T2
  The Strengths and Difficulties Questionnaire (SDQ) is a 25-item emotional and behavioural screening questionnaire for children and young people. The version for the parents of 4-17-year-olds will be used. Each item is rated on a 3-point scale ('not true', 'somewhat true', 'certainly true'). The Chinese parent version showed good validity and reliability (Cronbach's alpha: 0.81).

OTHER OUTCOMES:
Train-the-trainer outcome | T1: Baseline, before the workshop; T2: Immediate after the workshop; T3: 10 months after baseline.
  Social workers' understanding of NVC will be assessed at TTT1-TTT3. Overall satisfaction with the workshops will be assessed during TTT2. Items are rated on a 5-point Likert scale (0 = strongly disagree to 5 = strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Grace Yuying Sun, Principal Investigator — Hong Kong Metropolitan University
Locations (1):
- The Jockey Club Institute of Healthcare of Hong Kong Metropolitan University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
We are not sharing individual participant data (IPD) due to privacy concerns and limitations in participant consent. Although the data is de-identified, there remains a risk of re-identification, and participants were not explicitly consented for public data sharing. Aggregate results will be made available through publications and presentations to ensure transparency.